CLINICAL TRIAL: NCT04816708
Title: A Self-directed Mobile Mindfulness Intervention to Address Distress and Burnout in Frontline Healthcare Workers
Acronym: LIFT-HCW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00107657
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Results first posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Emotional Distress; Burnout, Professional; Stress, Job; Anxiety; Depressive Symptoms
Keywords: Emotional distress; COVID-19; Burnout
MeSH Terms: conditions — Burnout, Professional; Occupational Stress; Anxiety Disorders; Depression; COVID-19; Burnout, Psychological

STUDY DESIGN:
Intervention Model Description: Single site, pilot randomized waitlist control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Intervention group (access to LIFT mindfulness app) (Active Comparator): Participants randomized to the intervention arm will be provided access to LIFT app's daily mobile mindfulness therapy for 30 days.
  Interventions: Behavioral: LIFT Mindfulness
- Arm 2: Control waitlist group (delayed access to LIFT mindfulness app) (No Intervention): Control participants will not receive access to the LIFT app daily mobile mindfulness therapy during study period. They may have access to LIFT app daily mobile mindfulness therapy after completion of the study period.

INTERVENTIONS:
Behavioral: LIFT Mindfulness — Mindfulness is a type of mind-body therapy that promotes a practice of non-judgmental awareness that can alleviate distress by uncoupling emotional reactions and habitual behavior from unpleasant symptoms, thoughts, and emotions. LIFT is a mobile mindfulness app which can assess levels of emotional distress via survey, and subsequently offer mindfulness content that has previously been used in ICU patients, where it was shown to reduce symptoms of depression, anxiety, and PTSD.
  Arms: Arm 1: Intervention group (access to LIFT mindfulness app)

SUMMARY:
This is a pilot randomized waitlist control trial assessing if the feasibility of using a mobile mindfulness app to treat emotional distress and burnout amongst nurses taking care of COVID-19 patients. This trial will help inform the study team if dissemination the intervention to a large number of nurses in a short time period is feasible, and if the intervention has evidence of a clinical impact.

DETAILED DESCRIPTION:
Emotional distress and burnout are common among health care workers, particularly among nurses. These burdens have been worsened due to the COVID-19 pandemic's imposition of substantial physical and psychological stressors as well as persistent worry about personal health. There are few effective therapies for healthcare workers' symptoms of distress, fewer still that can be easily scaled, and most require face-to-face contact which is discouraged during a pandemic.

Mindfulness is a type of mind-body therapy that promotes a practice of non-judgmental awareness that can alleviate distress by uncoupling emotional reactions and habitual behavior from unpleasant symptoms, thoughts, and emotions. LIFT is a mobile mindfulness app which can assess levels of emotional distress via survey, and subsequently offer mindfulness content.

The LIFT-Healthcare Worker pilot randomized control trial (RCT) seeks to address those unmet needs. The trial will explore the feasibility and impact of the LIFT mobile app in relieving symptoms of emotional distress among nurses directly caring for COVID-19 patients in the Duke University Health System.

Target enrollment is for up to 200 participants. After signing consent, participants will be randomized via the LIFT app in a 2:1 (intervention:control) fashion into two arms:

1. Arm 1: Intervention group (access to LIFT mindfulness app)
2. Arm 2: Control waitlist group (delayed access to LIFT app)

Aim 1, which is to determine the feasibility of using the LIFT app among nurses directly caring for COVID-19 patients, will be assessed via the app which tracks user fidelity and adherence, and the use of an interactive dashboard for administrative users (i.e., study team) to track individual participant use. An open ended narrative question at 1 month will also help provide guidance for improving usability in future studies, as will directed telephone interviews with participants with high and low app.

Aim 2, which is to assess evidence of clinical impact of LIFT compared to control among nurses directly caring for COVID-19 patients at 1 month, will be assessed by comparing changes in the Patient Health Questionnaire-9 (PHQ-9), General Anxiety Disorder -7 (GAD-7) questionnaire, the Maslach Burnout Index (MBI), and Perceived Stress Scale 4 (PSS-4) over the study duration (1 month) between intervention and usual care groups.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 years of age
2. Currently working as a nurse in an adult COVID unit at Duke University Hospital
3. English Fluency

Exclusion Criteria:

1. Lack of access to either reliable smartphone with cellular data plan or home internet access.
2. Anticipation of leaving current position in ≤30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cox, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pratt EH, Hall L, Jennings C, Olsen MK, Jan A, Parish A, Porter LS, Cox CE. Mobile Mindfulness for Psychological Distress and Burnout among Frontline COVID-19 Nurses: A Pilot Randomized Trial. Ann Am Thorac Soc. 2023 Oct;20(10):1475-1482. doi: 10.1513/AnnalsATS.202301-025OC. PMID 37289650

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from May 19, 2021 - December 15, 2021 via flyer and/or email which contained QR code and/or URL to download app. Flyers were distributed in eligible hospital units, and emails were sent to listservs for nurses working in eligible units.
Period: Overall Study
Arm/Group | Arm 1: Intervention Group (Access to LIFT Mindfulness App) | Arm 2: Control Waitlist Group (Delayed Access to LIFT Mindfulness App)
Started | 69 | 33
Completed | 59 | 29
Not Completed | 10 | 4
Not completed — Lost to Follow-up | 10 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Intervention Group (Access to LIFT Mindfulness App) | Arm 2: Control Waitlist Group (Delayed Access to LIFT Mindfulness App) | Total
Number analyzed (Participants) | 69 | 33 | 102
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27 [25 to 32] | 25 [25 to 35] | 26.5 [25 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 31 | 96
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 1 | 8
  Not Hispanic or Latino | 62 | 32 | 94
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 60 | 27 | 87
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 69 | 33 | 102

OUTCOME MEASURES:

1. Primary Outcome: Intervention Completion
Description: The percentage of participants who complete all 4 weeks of the intervention, a measure of feasibility.
Time Frame: 30 days post randomization
Population: Not applicable to the control group.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Intervention Group (Access to LIFT Mindfulness App) | Arm 2: Control Waitlist Group (Delayed Access to LIFT Mindfulness App)
Number analyzed (Participants) | 69 | 0
percentage of participants | 28 |

2. Primary Outcome: Sessions Completed
Description: Number of daily mindfulness sessions completed by participants in intervention arm, a measure of feasibility.
Time Frame: 30 days post-randomization
Population: Not applicable to the control group.
Measure: Median (Inter-Quartile Range); unit: sessions per day
Arm/Group | Arm 1: Intervention Group (Access to LIFT Mindfulness App) | Arm 2: Control Waitlist Group (Delayed Access to LIFT Mindfulness App)
Number analyzed (Participants) | 69 | 0
sessions per day | 3 [1 to 17] |

3. Primary Outcome: Survey Completion at Baseline
Description: The percentage of patients who complete surveys at baseline, a measure of feasibility.
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Intervention Group (Access to LIFT Mindfulness App) | Arm 2: Control Waitlist Group (Delayed Access to LIFT Mindfulness App)
Number analyzed (Participants) | 69 | 33
percentage of participants | 100 | 100

4. Primary Outcome: Survey Completion at 1 Month
Description: The percentage of patients who complete surveys at 1 month, a measure of feasibility.
Time Frame: 30 days post randomization
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Intervention Group (Access to LIFT Mindfulness App) | Arm 2: Control Waitlist Group (Delayed Access to LIFT Mindfulness App)
Number analyzed (Participants) | 69 | 33
percentage of participants | 86 | 88

5. Secondary Outcome: Change in Patient Health Questionnaire-9 Item Scale (PHQ-9)
Description: Depression symptoms. Scores range from 0 (better) to 27 (worse).
Time Frame: Baseline to 30 days post-randomization
Population: Data not collected on 14 participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1: Intervention Group (Access to LIFT Mindfulness App) | Arm 2: Control Waitlist Group (Delayed Access to LIFT Mindfulness App)
Number analyzed (Participants) | 59 | 29
score on a scale | -2.94 [-4.07 to -1.82] | -0.74 [-2.27 to 0.80]

6. Secondary Outcome: Change in Generalized Anxiety Disorder 7-item Scale (GAD-7)
Description: Anxiety symptoms. Scores range from 0 (better) to 21 (worse).
Time Frame: Baseline to 30 days post-randomization
Population: Data not collected on 14 participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1: Intervention Group (Access to LIFT Mindfulness App) | Arm 2: Control Waitlist Group (Delayed Access to LIFT Mindfulness App)
Number analyzed (Participants) | 59 | 29
score on a scale | -2.91 [-3.31 to -1.07] | -0.79 [-2.29 to 0.71]

7. Secondary Outcome: Change in Perceived Stress Scale (PSS-4)
Description: Stress symptoms. Scores range from 0 (better) to 16 (worse).
Time Frame: Baseline to 30 days post-randomization
Population: Data not collected on 14 participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1: Intervention Group (Access to LIFT Mindfulness App) | Arm 2: Control Waitlist Group (Delayed Access to LIFT Mindfulness App)
Number analyzed (Participants) | 59 | 29
score on a scale | -0.65 [-1.27 to -0.02] | -0.97 [-1.80 to -0.15]

8. Secondary Outcome: Change in Maslach Burnout Index (MBI) - Emotional Exhaustion
Description: All MBI items are scored using a 7 level frequency ratings from "never" to "daily." The MBI has three component scales: emotional exhaustion (9 items), depersonalization (5 items) and personal achievement (8 items). Each scale measures its own unique dimension of burnout. Reported here is the emotional exhaustion component, which has a score range of 0-54, where a higher score indicates greater emotional exhaustion (indicative of burnout).
Time Frame: Baseline to 30 days post-randomization
Population: Data not collected on 14 participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1: Intervention Group (Access to LIFT Mindfulness App) | Arm 2: Control Waitlist Group (Delayed Access to LIFT Mindfulness App)
Number analyzed (Participants) | 59 | 29
score on a scale | -3.51 [-5.64 to -1.39] | -2.19 [-5.14 to 0.75]

9. Secondary Outcome: Change in Maslach Burnout Index (MBI) - Depersonalization
Description: All MBI items are scored using a 7 level frequency ratings from "never" to "daily." The MBI has three component scales: emotional exhaustion (9 items), depersonalization (5 items) and personal achievement (8 items). Each scale measures its own unique dimension of burnout. Reported here is the depersonalization component, which has a score range of 0-30, where a higher score indicates greater depersonalization (indicative of burnout).
Time Frame: Baseline to 30 days post-randomization
Population: Data not collected on 14 participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1: Intervention Group (Access to LIFT Mindfulness App) | Arm 2: Control Waitlist Group (Delayed Access to LIFT Mindfulness App)
Number analyzed (Participants) | 59 | 29
score on a scale | -0.29 [-1.19 to 0.61] | -1.89 [-3.11 to -0.66]

10. Secondary Outcome: Change in Maslach Burnout Index (MBI) - Personal Accomplishment
Description: All MBI items are scored using a 7 level frequency ratings from "never" to "daily." The MBI has three component scales: emotional exhaustion (9 items), depersonalization (5 items) and personal achievement (8 items). Each scale measures its own unique dimension of burnout. Reported here is the personal achievement component, which has a score range of 0-30, where a lower score indicates less sense of personal achievement (indicative of burnout).
Time Frame: Baseline to 30 days post-randomization
Population: Data not collected on 14 participants.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1: Intervention Group (Access to LIFT Mindfulness App) | Arm 2: Control Waitlist Group (Delayed Access to LIFT Mindfulness App)
Number analyzed (Participants) | 59 | 29
score on a scale | 0.23 [-1.11 to 1.57] | -0.63 [-2.49 to 1.22]

ADVERSE EVENTS:
Time Frame: Up to 30 days post-randomization
Arm/Group | Arm 1: Intervention Group (Access to LIFT Mindfulness App) | Arm 2: Control Waitlist Group (Delayed Access to LIFT Mindfulness App)
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/29
Other Adverse Events (participants affected / at risk) | 1/59 | 0/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Intervention Group (Access to LIFT Mindfulness App) (N=59) | Arm 2: Control Waitlist Group (Delayed Access to LIFT Mindfulness App) (N=29)
Suicidal Ideation (Psychiatric disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT04816708/Prot_SAP_000.pdf